CLINICAL TRIAL: NCT06542445
Title: The Safety and Efficacy of Treatment With Cannabidiol (CBD) Oil Enriched With Terpenes, Devoid of THC, in Children Diagnosed With ADHD
Brief Title: The Safety and Efficacy of Terpene-enriched Cannabidiol (CBD) Oil in ADHD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bazelet Nehushtan LtD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASF-0243-22
Record Dates: First submitted 2024-07-31; First posted 2024-08-07 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: Cannabidiol; Terpenes; Medical Cannabis; Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Terpenes

STUDY DESIGN:
Intervention Model Description: Each participant will be randomly assigned to receive either the terpene-enriched CBD oil or a placebo for 5 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All blinded except dispensing pharmacist.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBD oil enriched with terpenes (Active Comparator): 24% CBD, terpenes, MCT oil.
  Interventions: Drug: Oral CBD oil enriched with terpenes
- Placebo oil (Placebo Comparator): fragrances and flavors, MCT oil.
  Interventions: Drug: Oral Placebo

INTERVENTIONS:
Drug: Oral CBD oil enriched with terpenes — Stage I dosing, increasing titration:
  days 1-2: 2.5 mg/kg BW/day; days 3-4: 5 mg/kg BW/day; day 5-7: 7.5 mg/kg BW/day; days 8-35: 10 mg/kg BW/day.
  Stage II dosing, increasing titration:
  days 36-37: 2.5 mg/kg BW/day; days 38-39: 5 mg/kg BW/day; day 40-42: 7.5 mg/kg BW/day; days 43-70:10 mg/kg BW/day.
  Arms: CBD oil enriched with terpenes
Drug: Oral Placebo — Oral placebo oil that is similar in appearance and taste to the CBD oil. Titration and dosing identical to those described for the CBD oil.
  Arms: Placebo oil

SUMMARY:
ADHD is the most frequent neurodevelopmental disorder in childhood. Symptoms often appear in preschool years, and most children (65-80%) continue to experience some ADHD-associated symptoms into adolescence and adulthood. The disorder is marked by age-inappropriate inattention, hyperactivity, and impulsivity. Drug treatments for ADHD include stimulants containing methylphenidate (like Ritalin and Concerta) or amphetamines (like Vyvanse). However, 30-35% of the patients do not respond well to these treatments, and stimulants may result with various side effects.

The use of medical cannabis increases; applied for expending medical conditions, with growing evidence for its beneficial effects. A study on ADHD adults treated by cannabinoids demonstrated improvements in hyperactivity and impulsivity.

The current study is aimed to examine the safety and efficacy of treating children diagnosed with ADHD with a CBD oil (devoid of THC), enriched with terpenes. Participants will be randomly assigned to receive either the enriched CBD oil or a placebo, for 5 weeks (Treatment, Stage I).

At the end of the treatment stage (I), an open-label stage will follow (II), wherein, all participants will receive the investigational product for an additional 5 weeks.

The investigators hypothesize that children treated with the enriched CBD oil (Treatment, Stage I) will show significantly higher improvement in hyperactivity and inattention scores, as compared with the placebo group.

DETAILED DESCRIPTION:
Screening phase:

Parents who are interested to take part in study, will contact the study team. Parents will be asked to provide documents attesting their child's medical status and forms required to process a medical cannabis prescription.

Visit 1 - Baseline:

* Participants and parents will sign an Informed Consent Form.
* Parents will complete questionnaires about the child's health, clinical history, medications, sleep, eating habits, and quality of life.
* Participants will be examined by a pediatrician, who will fill out a physical examination report, including height, weight and blood pressure, and will conduct an urine test.
* Participants will conduct a TOVA (Test of Variables of Attention) test, and answer a CBCL (Child Behavior Checklist) questionnaire.
* Parents and teachers will complete the Conners questionnaires (sent during the screening phase. Conners questionnaires may be filled out prior to Visit 1, but no longer than two weeks prior to Visit 1).
* Participants and parents will receive the study drug/placebo and usage instructions.

Treatment using the study drug (Stage I) will be initiated following Visit 1, according to a schedule set by the study team.

Follow-up 1:

The study team will contact the parents via a phone call two weeks (±2 days) after initiation of stage I. Parents will answer questions regarding general health and side effects.

Visit 2 -at the end of Stage I:

* Five weeks (±3 days) after initiation of stage I.
* Participants and parents will undergo and fill out the same set of examinations and questionnaires as in Visit 1.
* All participants will receive new bottles of the investigational product - the CBD oil enriched with terpenes (open label, Stage II).

Follow-up 2:

• The study team will contact the parents via a phone call two weeks (±2 days) after initiation of Stage II. Parents will answer questions regarding general health and side effects.

Visit 3 - at the end of Stage II:

* Five weeks (±3 days) after initiation of stage II.
* Participants and parents will undergo and fill out the same set of examinations and questionnaires as in Visit 1, excluding the TOVA test.
* Study drugs' bottles and cannabis use prescription will be returned to the study team.

ELIGIBILITY:
Inclusion Criteria:

1. Children/adolescents aged 6-18 diagnosed with ADHD as per DSM-V by a neurologist, psychiatrist or other specialist.
2. Willing/able to arrive to all the necessary visits as per study protocol.

Exclusion Criteria:

1. Participants who used ADHD conventional medications in the month before starting the study or intend to do so during the study.
2. Participants who used benzodiazepines or first-generation antihistamines in the week before starting the study or other drugs which may interfere with the study as per PI opinion.
3. Participants suffering from neurological or psychiatric diseases.
4. Participants suffering from neoplastic diseases.
5. Participants with syndromes or metabolic diseases.
6. Participants with a significant clinic diagnosis which may interfere with the study. May be included later on as per PI opinion.
7. Pregnant or breastfeeding adolescents.
8. Sexually active female adolescents who are unwilling to use contraceptives.
9. Participants that in the PI opinion will not comply with the protocol in a way that will harm the study (for ex.: not using contraceptives.)
10. Participants with less than 18 kg or more than 90 kg weight.
11. Participants with BMI lower than 18 or higher than 29.9.
12. Participants engaged in another clinical study which includes a medicine.
13. Participants engaged in another study regarding ADHD treatment of any kind.
14. Participants using alcohol or drugs.
15. Past or present use of Cannabis, including medical cannabis

Criteria for early termination:

1. Use of another medication for ADHD during the study.
2. Use of a medication from the exclusion criteria list during the study.
3. Use of alcohol or drugs during the study.
4. Participants who got pregnant during the study.
5. Participants who split the first visit and did not arrive to the second part of the first visit after a maximum of 28 days.
6. Participants who did not start the treatment during the 14 days from receiving the drug.
7. Non -compliant participants.

Criteria for exchange:

1. PI may exchange participants that quit, if they did not start treatment for new participants.
2. PI may recruit again participants who quit after a new full recruitment process.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2026-08-22 (Estimated); Study Completion 2026-09-22 (Estimated)

PRIMARY OUTCOMES:
Improvement in hyperactivity sub-score of the Conners' Parent Questionnaire, as compared with baseline. | 5 weeks (Visit 1 to Visit 2)
  Conners' Parent Rating Scale
Improvement in inattentiveness sub-score of the Conners' Parent Questionnaire, as compared with baseline. | 5 weeks (Visit 1 to Visit 2)
  Conners' Parent Rating Scale

SECONDARY OUTCOMES:
Improvement in Conners' Parent Questionnaire - Total score, as compared with baseline. | 5 weeks (Visit 1 to Visit 2)
  Conners' Parent Rating Scale
Improvement in hyperactivity sub-score of the TOVA test, as compared with baseline. | 5 weeks (Visit 1 to Visit 2)
  Computerized visual T.O.V.A
Improvement in inattentiveness sub-score of the TOVA test, as compared with baseline. | 5 weeks (Visit 1 to Visit 2)
  Computerized visual T.O.V.A
Improvement in TOVA test - Total score, as compared with baseline. | 5 weeks (Visit 1 to Visit 2)
  Computerized visual T.O.V.A
Improvement in hyperactivity sub-score of the Conners' Teacher Questionnaire, as compared with baseline. | 5 weeks (Visit 1 to Visit 2)
  Conners' Teacher Rating Scale
Improvement in inattentiveness sub-score of the Conners' Teacher Questionnaire, as compared with baseline | 5 weeks (Visit 1 to Visit 2)
  Conners' Teacher Rating Scale
Improvement in Conners' Teacher Questionnaire - Total score, as compared with baseline. | 5 weeks (Visit 1 to Visit 2)
  Conners' Teacher Rating Scale
Improvement in the scores of CBCL questionnaire, as compared with baseline. | 5 weeks (Visit 1 to Visit 2)
  Child Behavior Checklist (CBCL)
Side effects are tolerable and transient. | 5 weeks (Visit 1 to Visit 2)
  Side effect questionnaire
The rate of drop-out will be similar in both groups. | 5 weeks (Visit 1 to Visit 2)
  Drop-outs will be recorded by the study stuff.

CONTACTS AND LOCATIONS:
Overall Officials: Matitiahu Berkovitch, MD, Principal Investigator — Shamir Medical Center, Zerifin, Israel
Locations (1):
- Shamir Medical Center, Ẕerifin, Israel